CLINICAL TRIAL: NCT07188740
Title: Metformin Inhibits DNMT3A Clonal Hematopoiesis in Acute Leukemia: A Single-Arm Clinical Study
Brief Title: Metformin Inhibits DNMT3A Clonal Hematopoiesis in Acute Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025104
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: DNMT3A Gene Mutation
Keywords: CHIP; acute leukemia; Metformin; DNMT3A
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin Treatment Arm (Experimental): Dosage: Start at 500 mg twice daily, titrate to 2000 mg/day (e.g., 500 mg three times daily or 1000 mg twice daily), based on tolerance.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Start at 500 mg twice daily, titrate to 2000 mg/day for 6 months

SUMMARY:
This is a prospective, single-arm clinical study evaluating the efficacy and safety of metformin in inhibiting DNMT3A R882-driven clonal hematopoiesis (CH) in patients with acute leukemia (AL) who are in remission and under follow-up. Patients with DNMT3A R882 mutation (VAF ≥5%) will receive oral metformin for 6 months, with dosage gradually increased to 2000 mg/day. The primary endpoint is the proportion of patients with effective decline in DNMT3A R882 mutation VAF at 6 months. Secondary endpoints include VAF decline at 3 months, relapse-free survival (RFS) at 6 and 12 months, overall survival (OS), cumulative incidence of relapse (CIR), cumulative remission-phase mortality, and adverse event rates. Planned enrollment: 30 participants.

DETAILED DESCRIPTION:
Clonal hematopoiesis (CHIP) involves hematopoietic stem cells (HSCs) acquiring mutations like DNMT3A R882, conferring a proliferative advantage and increasing risks of hematologic malignancies and inflammatory diseases. No effective interventions exist currently. Preclinical studies show that DNMT3A R882 mutations enhance mitochondrial respiration and oxidative phosphorylation (OXPHOS) in hematopoietic stem/progenitor cells (HSPCs), which is essential for their competitive advantage. Metformin, at clinical doses, inhibits the electron transport chain (ETC) complex I, reducing OXPHOS and selectively diminishing the advantage of mutant HSPCs. Mechanisms include restoring epigenetic stability by elevating methylation potential (SAM/SAH ratio), reversing hypomethylation in differential methylation regions (DMRs), and normalizing H3K27me3 histone modifications.

In mouse and humanized models, metformin suppresses clonal expansion of DNMT3A R882 mutant cells. Based on metformin's 60-year safety profile in diabetes treatment, this study tests its potential in AL patients with persistent DNMT3A R882 CH post-remission. Metformin may reduce risks like secondary tumors and diabetes in these patients.

Study intervention: Oral metformin starting at 500 mg twice daily, titrated to 500 mg three times daily or 1000 mg twice daily (or maximum tolerated dose), up to 2000 mg/day, taken with meals for 6 months.

Efficacy assessment: Next-generation sequencing (NGS) for DNMT3A R882 VAF at 0, 3, and 6 months.

* Major response: For VAF >20%, absolute decline ≥10%; for VAF ≤20%, relative decline ≥50%.
* Partial response: For VAF >20%, absolute decline 5-10%; for VAF ≤20%, relative decline 25-50%.

Safety monitoring: Close monitoring of liver/kidney function, especially in patients ≥60 years or with renal impairment, due to lactic acidosis risk.

Data management uses electronic case report forms (eCRF). Statistical analysis includes intention-to-treat (ITT) and per-protocol (PP) sets, with Kaplan-Meier for survival, t-tests, Wilcoxon rank-sum, chi-square, and Cox proportional hazards models.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute leukemia based on bone marrow morphology, immunology, and genetics, per WHO 2022 or ICC criteria.
* Patients in complete remission follow-up phase with DNMT3A R882 mutation clonal hematopoiesis, VAF ≥5%.
* Age ≥14 years, any gender
* Laboratory requirements (within 7 days before treatment):

  * Total bilirubin ≤1.5 × upper limit of normal (ULN) for age.
  * AST and ALT ≤2.5 × ULN for age.
  * Serum creatinine <2 × ULN for age.
  * Cardiac enzymes <2 × ULN for age.
  * Ejection fraction within normal range by echocardiogram (ECHO).
* Signed informed consent: By patient (≥18 years) or legal guardian/relative (<18 years or if beneficial for condition).

Exclusion Criteria:

* Patients with diabetes receiving other medications
* Known allergy to metformin
* Deemed unsuitable by investigator

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
DNMT3A R882 Mutation VAF at 6 Months | up to 6 months
  Effective decline defined as: For baseline VAF >20%, absolute decline ≥10%; for VAF ≤20%, relative decline ≥50%. Measured via NGS.

SECONDARY OUTCOMES:
DNMT3A R882 Mutation VAF at 3 Months | up to 3 months
  Same criteria as primary endpoint. Measured via NGS
Relapse-Free Survival (RFS) Rate at 6 Months | up to 6 months
  Proportion of patients without relapse
Relapse-Free Survival (RFS) Rate at 12 Months | up to 12 months
  Proportion of patients without relapse
Overall Survival (OS) Rate | Up to 12 months
  Proportion of patients alive
Cumulative Incidence of Relapse (CIR) | Up to 12 months
  Cumulative rate of relapse events
Cumulative Remission-Phase Mortality Rate | Up to 12 months
  Cumulative rate of deaths during remission